CLINICAL TRIAL: NCT00582387
Title: Pilot Study: Genetic Susceptibility to Tumor Recurrence and Progression in Patients With Non-Muscle Invasive Bladder Cancer
Brief Title: Genetic Susceptibility to Tumor Recurrence and Progression in Patients With Non-Muscle Invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-011
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Cancer; Urinary Cancer; Nonmuscle Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine and tissue

GROUPS / COHORTS (1):
- nonmuscle invasive bladder cancer: This is a hospital-based cohort study in which subjects with non-muscle invasive bladder cancer diagnosed within the previous 12 months will be evaluated to determine whether candidate genetic variants in patients with superficial bladder cancer can predict the risk of disease recurrence and/or progression, with the goal of modifying surveillance schedules as a function of predicted risk of recurrence or progression. All patients will be treated according to the treatment plan as outlined by their attending physician. The study will not require any deviation from the planned usual treatment.
  Interventions: Genetic: specimen samples; Behavioral: questionnaires

INTERVENTIONS:
Genetic: specimen samples — blood, urine and tissue
Behavioral: questionnaires

SUMMARY:
The purpose of the study is to see if we will be more able to tell what the risk is for bladder cancer to reoccur or worsen when genetics and risk factors are examined along with the stage and grade of the tumor. Superficial bladder cancer is a cancer that does not grow into the muscle layer of the bladder wall. Even though it is a superficial cancer, this type of cancer tends to come back after being treated and is often more aggressive when it returns. We already know, that the "stage" or how deeply the tumor grows into the bladder wall and the "grade" or how fast the tumor grows affect whether the tumor will come back or get worse over time. Now we use information about the stage and grade of your tumor to decide how to treat the tumor and how often you should be checked after the treatment is over. However, this has not been very reliable, because each person has unique genetic characteristics and other factors that are likely to affect what happens to the tumor over time. For instance, we know the risk for developing a cancer may be affected by your surroundings and other factors such as what you eat, the type of habits you have such as smoking, and the type of job you have, but not everyone exposed to the same risk factors gets a cancer. We believe this is due to unique genetic characteristics in each person which may help their body fight cancer.

DETAILED DESCRIPTION:
This is a hospital based cohort study where subjects diagnosed within twelve months with nonmuscle invasive bladder cancer will be evaluated to determine whether candidate genetic variants are associated with the risk of recurrence and progression. Known tumor variables will be stratified and correlated with markers. The long term goal is to estimate the predicted risk of recurrence or progression well enough to modify surveillance schedules. Since 40% of superficial bladder cancer patients will never recur or progress, these individuals could return less frequently for followup, saving costs and discomfort. All patients will receive usual care and be followed to determine rates of recurrence and progression of the disease. Each subject will donate 30 ml of blood for extraction of genomic DNA and isolation of lymphocytes to assess DNA damage/repair function. In addition, each subject who undergoes a transurethral resection of the bladder (TURB) and/or random bladder biopsies as part of his/her usual care will donate urothelial cells from the random bladder biopsies for analyses of DNA damage/repair function. The DNA repair capacity of lymphocytes will be correlated with that of normal bladder tissue to evaluate the use of lymphocytes as a surrogate marker. When bladder biopsy tissue is not available, urothelial cells will be obtained from a cystoscopic or catheterized bladder lavage.

ELIGIBILITY:
Inclusion Criteria:

* They have been diagnosed with a primary nonmuscle invasive bladder cancer within the previous 12 months.
* They speak English or a language for which we have a translated consent form
* They understand and agree to sign informed consent
* They agree to donate a 30ml blood sample
* They agree to give us a bladder tissue sample as part of normal clinical procedures (three 3mm cold cup bladder biopsies or urothelial cells by bladder lavage)
* They agree to complete the study questionnaires
* They agree to have their pathology information reviewed. This could include biopsy specimens.
* All subjects must be age 21 or older

Exclusion Criteria:

* Age less than 21 years
* History of other cancer diagnosis excluding nonmelanoma skin cancers
* History of muscle invasive bladder cancer
* Initial diagnosis more than 12 months from entry date into study
* History of prior intravenous chemotherapy or radiation therapy
* Bladder histology other than transitional cell cancer and its variants.
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology clinic
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2004-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluate genetic variants (in the DNA repair genes, cell cycle genes, and detoxifying genes) and their association with recurrence and progression in early stage bladder cancer. | conclusion of study

SECONDARY OUTCOMES:
Compare the DNA damage/repair capacity with the genetic variants. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Donat, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org